CLINICAL TRIAL: NCT00485160
Title: Comparison of Intravenous Ibuprofen vs. Continuous Indomethacin in the Treatment of Patent Ductus Arteriosus
Brief Title: Ibuprofen vs. Continuous Indomethacin in the Treatment of PDA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Cathy Hammerman, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: chammerman2
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2007-06

CONDITIONS: Patent Ductus Arteriosus
Keywords: Patent Ductus Arteriosus; Indomethacin; Ibuprofen; Renal effects
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Continuous indomethacin
Drug: ibuprofen

SUMMARY:
The purpose of this study is to determine whether closure of the PDA in premature neonates using IV ibuprofen vs continuous IV indomethacin has different side effects, eg. effects on renal function, on blood flow velocity in the superior mesenteric artery, the anterior cerebral artery, and the renal artery.

DETAILED DESCRIPTION:
Despite the fact that ibuprofen appears to minimize the renal side effects seen following bolus indomethacin, other concerns regarding both short and long-term safety remain. Indomethacin, on the other hand, has been used to treat premature neonates for many years. Other than transient vasoconstrictive effects, no significant toxicity has been noted. Thus, if we were to be able to eliminate the differential renal effects, indomethacin would remain, for many, the therapy of choice for the premature neonate with a persistent PDA. We hypothesized that continuous administration of indomethacin would provide this option. Ibuprofen therapy has not, to date, been compared with indomethacin administered by continuous infusion. Hence, in the current study we attempted to determine whether continuous indomethacin administration could potentially offer the same advantages as ibuprofen in treating PDA, specifically in terms of mitigation of renal side effects. Specifically, our primary objective was to show no differences in urine output and/or in serum creatinine between the treatment groups. As a secondary objective, we aimed to show no other potentially vascular-mediated clinical differences, eg. Necrotizing enterocolitis (NEC), intraventricular hemorrhage (IVH), retinopathy of prematurity (ROP) and on bilirubin albumin binding between the groups.

B-type natriuretic peptide (BNP) is released by ventricular myocytes in response to ventricular volume load. It, in turn, mediates vasodilation, natriuresis and diuresis. Serum BNP levels have been shown to be clinically useful in differentiating between respiratory and cardiac disease, in monitoring heart failure therapies and in serving as early diagnostic biomarkers of ductal patency in premature neonates. As secondary objectives we intend to determine whether a decrease in BNP levels would be an equally reliable indicator of therapeutic efficacy in infants treated with ibuprofen as with indomethacin.In addition we will look at comparative effects on other vascular beds which might mediate long term side effects described above.

ELIGIBILITY:
Inclusion Criteria:

* < 1500 gm birth weight with PDA confirmed by echocardiography

Exclusion Criteria:

* Additional congenital heart lesions
* Significant congenital malformations
* Documented infection
* Thrombocytopenia (<60,000)
* IVH grade 4

Ages: 36 Hours to 3 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2002-02; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To show no differences in urine output and/or in serum creatinine between the treatment groups | Up to one day after completion of therapy

SECONDARY OUTCOMES:
To show no other clinical differences, eg. NEC, IVH or ROP between the groups; to study doppler flow velocities to these areas; to correlate with BNP levels. | Until end of primary hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Hammerman, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel